CLINICAL TRIAL: NCT03337009
Title: The Impact of a Web-Based Naloxone Intervention Under Standing Orders to Patients Prescribed Chronic Opioid Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CO-16-2405-01; 1R01DA042059 (NIH)
Record Dates: First submitted 2017-10-16; First posted 2017-11-08 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Overdose; Risk Behavior
Keywords: Opioid antagonist; Naloxone; Opioids; Web-based intervention
MeSH Terms: conditions — Drug Overdose; Risk-Taking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxone Navigator (Experimental): Targeted, web-based animated video (Naloxone Navigator [NN]):
  This arm is a web-based intervention targeted to patients receiving chronic opioid therapy identified in the electronic health record. Participants in this arm have access to naloxone under standing orders from the pharmacy or with a prescription from their providers.
  Interventions: Behavioral: Naloxone Navigator (NN)
- Usual Care (No Intervention): Participants in the usual care arm will receive usual care from their health plan, pharmacy and clinicians. As part of usual care, participants can access naloxone through physician prescription or standing orders.

INTERVENTIONS:
Behavioral: Naloxone Navigator (NN) — Patients prescribed chronic opioid therapy will be identified and recruited to enroll in the study. Patients randomized to receive the web-based animated video (Naloxone Navigator) will be sent a link to the video after enrollment. The web-based, animated video provides education on what is an opioid overdose, how to prevent it, how to recognize an overdose, and how to respond with naloxone. This video also encourages patients to pick up naloxone from a pharmacy under a standing order.
  Arms: Naloxone Navigator

SUMMARY:
In the setting of naloxone standing orders, this study will assess the impact of a targeted, web-based overdose prevention and naloxone intervention for patients prescribed chronic opioid therapy. Outcomes are changes in opioid risk behaviors, naloxone uptake, and knowledge about overdose and naloxone.

DETAILED DESCRIPTION:
This is a patient level randomized study of a targeted, web-based overdose prevention and naloxone intervention for patients prescribed chronic opioid therapy. This study will be conducted in a health system which has implemented naloxone standing orders. Adults prescribed chronic opioid therapy will be identified in the electronic health record, outreached, and recruited for participation. Once enrolled, participants will be randomized to usual care or the intervention. The web-based intervention is an animated video which provides education on what is an opioid overdose, how to prevent and recognize an opioid overdose, and how to respond with naloxone. This video also encourages patients to pick up naloxone from a pharmacy under standing orders. Participants will be given knowledge and risk surveys over the follow-up. The primary outcome is opioid risk behavior. Secondary outcomes include knowledge about overdose and naloxone, substance use, and pain intensity. Patients will also be followed in the electronic health record for naloxone dispensings, changes in opioid dose, aberrant urine toxicology results, and overdose events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Prescribed chronic opioid therapy
* Have a health plan which covers the formulation of naloxone available at the pharmacy they received their opioid prescriptions from.

Exclusion Criteria:

* Non-English speaking, hospice enrollment, do-not-resuscitate order, no internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Opioid-Related Risk Behavior | Change from baseline to 4-6 months, and 8-12 months
  Risk behavior will be assessed using the Opioid-Related Behaviors in Treatment (ORBIT) scale. The ORBIT is a scale used to identify recent risk behavior among patients receiving chronic opioid therapy. Scores on the single scale range from 0-40, with lower values representing less risk behavior.

SECONDARY OUTCOMES:
Overdose and Naloxone Knowledge | Baseline post-intervention and sustained effects at 4-6 and 8-12 months
  Patient knowledge of overdose and naloxone will be measured using survey items adapted from the Opioid Overdose Knowledge Scale (OOKS). The OOKS is a scale measuring knowledge of overdose risks, warning signs, steps to address the overdose and appropriate use of naloxone. The investigators have adapted it to be specific to prescription opioids. The modified-OOKS is scored on a scale of 0-28, with higher values representing greater knowledge about overdose and naloxone.
Rate of Naloxone Dispensings | Baseline to 12 months
  Pharmacy or insurance claims databases will be used to identify naloxone dispensings in the outpatient setting.
Patient reported naloxone pick-up | Baseline to 12 months
  Patient surveys will be used to identify naloxone dispensings in the outpatient setting.
Change in opioid dose | Baseline to 12 months
  Using pharmacy or insurance claims data, the investigators will calculate changes in the milligrams morphine equivalent dose.
Change in Drug Use Risk Behavior | Change from baseline to 4-6 months, and 8-12 months
  Drug Use Risk Behavior will be assessed using question 2 of the validated National Institutes on Drug Abuse-Modified Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) scale version 2.0. Scores on the single scale range from 0-60, with lower values representing less drug use risk behavior.
Change in Hazardous Drinking and Alcohol Use Disorders | Change from baseline to 4-6 months, and 8-12 months
  Alcohol Use Risk Behavior will be assessed using the validated Alcohol Use Disorders Identification Test--Consumption (AUDIT-C) scale. AUDIT-C is a screener used to identify patients with alcohol use disorders or hazardous drinking behavior. The AUDIT-C is scored on a scale of 0-12. The higher the score, the more likely it is that the patient's drinking is affecting his or her safety.

OTHER OUTCOMES:
Change in Pain Intensity | Change from baseline to 4-6 months, and 8-12 months
  Pain intensity will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS Scale v1.0 - Pain Intensity 3a. The PROMIS Pain Intensity instrument is scored on a scale of 3-15. A higher score represents greater pain intensity.
Rate of Opioid Overdose | Baseline to 12 months
  Overdoses will be assessed using self-report, electronic health record data and death records.
Rate of Aberrant Urine Toxicology Screens | Baseline to 12 months
  Urine toxicology screen results found in laboratory databases will be used to measure opioid medication diversion and drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Binswanger, MD, Principal Investigator — Kaiser Permanente; Jason Glanz, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators interested in using the data from this study must submit a written request. Requests must address regulatory and compliance requirements for data usage. Investigators must outline the necessary resources required to support their data request, including personnel and infrastructure. The original study team will evaluate each request based on scientific merit, ethical considerations, and alignment with the original study's objectives.
  Deidentified survey and electronic health record (EHR) data will be shared with investigators upon approval of written request. Investigators are responsible for obtaining necessary approvals and adhering to relevant laws and regulations and will be required to sign a Data Use Agreement (DUA) outlining the terms and conditions of data usage. The data sharing period is limited to three years following the publication of the primary study. The Naloxone Navigator video is available upon request; please send an email to: jason.m.glanz@kp.org.
Supporting Information: Study Protocol
Time Frame: 3 years following the publication of the primary study
Access Criteria: See plan description

REFERENCES:
- [Derived] Glanz JM, Mueller SR, Narwaney KJ, Wagner N, Xu S, Kraus C, Wain K, Botts S, Binswanger IA. Effectiveness of direct patient outreach with a narrative naloxone and overdose prevention video to patients prescribed long-term opioid therapy in the USA: the Naloxone Navigator randomised clinical trial. BMJ Public Health. 2024 Jul;2(1):e000725. doi: 10.1136/bmjph-2023-000725. Epub 2024 Jul 8. PMID 39421268